CLINICAL TRIAL: NCT00549991
Title: Fine Mapping of Hypertension Genes Detected by Admixture Mapping in the FBPP
Brief Title: Analyzing Genes That May Increase the Risk of Developing High Blood Pressure
Status: Completed | Type: Observational
Sponsor: Case Western Reserve University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1415; R01HL086718 (NIH)
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
High blood pressure is one of the most common health problems in the United States. Genetic variations may cause some people to be more susceptible to developing high blood pressure. This study will identify variations in genes known to play a part in the development of high blood pressure.

DETAILED DESCRIPTION:
High blood pressure affects nearly one third of all individuals in the United States. It is especially common in African Americans, with more than 40% of African Americans diagnosed with this condition. High blood pressure usually develops earlier in life and is more severe in African Americans than in other racial or ethnic groups. Many factors can cause high blood pressure, including stress, diet, diabetes, kidney disease, or obesity. Previous studies have also shown that genetic variations on two regions of chromosomes 6 and 21 may predispose some people to develop high blood pressure. Admixture mapping is a type of genetic analysis that aims to identify disease-causing genetic variations across different populations of people. Using admixture mapping, this study will examine previously collected genetic samples from African American participants in the Family Blood Pressure Program (FBPP) study and from African American, Mexican American, Nigerian, and Jamaican participants enrolled in other clinical studies. Study researchers will analyze the samples to identify and characterize genetic variations that are associated with an increased risk of high blood pressure in the African American population, as well as other racial and ethnic groups.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the FBPP study (African American [800 people with high blood pressure and 800 control group participants] and Mexican American participants)
* Participated in the American Family Study (African American participants)
* Participated in the Phenotyping Study (African American, Nigerian, and Jamaican participants)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Previously collected genetic samples from African American participants in the Family Blood Pressure Program (FBPP) study and from African American, Mexican American, Nigerian, and Jamaican participants enrolled in other clinical studies will be examined.
Sampling Method: Probability Sample
Enrollment: 8687 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Genetic variations | Measured through admixture mapping genetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhu, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States